CLINICAL TRIAL: NCT06207084
Title: Precision-based Teleexercise Trial to Increase Adherence in People With Disabilities
Brief Title: The Fit With Us Study
Acronym: FITWITHUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300011762; 90REGE0019 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Mobility Limitations; Disability Physical; Telehealth; Health Coaching; Physical Activity; Behavior, Health; eHealth; Health Literacy; Self Efficacy; Fatigue; Usability; Predictive Model
Keywords: telehealth; health coaching; disability
MeSH Terms: conditions — Mobility Limitation; Motor Activity; Health Behavior; Fatigue

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomization Model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- asynchronous exercise responder (Experimental): Individuals only receiving asynchronous exercise content and are responding
  Interventions: Behavioral: asynchronous content only
- Asynchronous exercise and health coaching responder (Experimental): Individuals receiving asynchronous exercise content and health coaching and are responding
  Interventions: Behavioral: Asynchronous content and health coaching and no live training
- Asynchronous exercise non-responder and 1 on 1 live training (Experimental): Individuals receiving asynchronous exercise content and are not responding. The are receiving 1 on 1 live exercise sessions.
  Interventions: Behavioral: asynchronous content only and 1 on 1 live training
- Asynchronous exercise and health coaching non-responder and 1 on 1 live training (Experimental): Individuals receiving asynchronous exercise content and health coaching and are not responding. The are receiving 1 on 1 live exercise sessions.
  Interventions: Behavioral: asynchronous content and health coaching and 1 on 1 training
- Asynchronous exercise non-responder and group live training (Experimental): Individuals receiving asynchronous exercise content and are not responding. The are receiving group live exercise sessions.
  Interventions: Behavioral: asynchronous content and group training
- Asynchronous exercise and health coaching non-responder and group live training (Experimental): Individuals receiving asynchronous exercise content and health coaching and are not responding. The are receiving group live exercise sessions.
  Interventions: Behavioral: Asynchronous content and health coaching and group training

INTERVENTIONS:
Behavioral: asynchronous content only — Receives asynchronous exercise content and no live training
  Arms: asynchronous exercise responder
Behavioral: Asynchronous content and health coaching and no live training — Receives asynchronous content, health coaching and no live training.
  Arms: Asynchronous exercise and health coaching responder
Behavioral: asynchronous content only and 1 on 1 live training — receives asynchronous content and live 1 on 1 training
  Arms: Asynchronous exercise non-responder and 1 on 1 live training
Behavioral: asynchronous content and health coaching and 1 on 1 training — receives asynchronous content, health coaching, and live training
  Arms: Asynchronous exercise and health coaching non-responder and 1 on 1 live training
Behavioral: asynchronous content and group training — receives asynchronous content and live group training
  Arms: Asynchronous exercise non-responder and group live training
Behavioral: Asynchronous content and health coaching and group training — receives asynchronous content, health coaching, and live group training
  Arms: Asynchronous exercise and health coaching non-responder and group live training

SUMMARY:
The purpose of this 32-week study is to use an innovative experimental design known as SMART (Sequential Multiple Assignment Randomized Trial), which will allow us to determine the best way to sequence the delivery of teleexercise (referred to as an adaptive intervention), combined with predictive analytics on participant adherence in a stepped program of physical activity interventions. All 257 participants will have access to a library of recorded video exercise content, and a weekly wellness article. Some participants will receive health coaching calls (1st randomization). Analytic data will be used to determine which participants are responding or not responding to the intervention. Participants not responding after 4 weeks will receive either live one-on-one or group exercise training (2nd randomization). After 8 weeks, the participant will receive only pre-recorded exercise content and articles for a 24-week maintenance phase (weeks 9-32). The study outcomes are: The effectiveness of the adaptive interventions; Exploring mediating and moderating variables; Sensitivity analysis of the predictive analytics.

DETAILED DESCRIPTION:
The proposed Sequential Multiple Assignment Randomized Trial (SMART) study seeks to develop an effective 32-week, resource sensitive strategy to improve physical activity levels in people with mobility impairments.

During the run-In period before the start of the intervention, interested individuals will consent to be part of the study. Once providing consent, Participants will respond to a baseline survey packet through REDCap. Participants must also complete a welcome call and set up an online account. Additionally, during the run-in period, the research team will ship an exercise tracker device, and an exercise band for the participant to wear during the intervention. The participant will receive an orientation call to assist them with using the website, setting up their exercise tracking device, and linking the device to the website. (see attached call outline)

After the run-in period, participants will be randomized into 1 of 2 groups: Asynchronous Exercise Program (AEP) and AEP + Smart Health Coaching (SHC). Finally, participants will be given access to the FitWithUs online platform, hosted on UAB servers, to access all the exercise content (exercise videos and articles). All participants will receive at least one new health and wellness article per week for eight weeks, and new exercise videos for 16 weeks.

The Adoption Phase will be split into two 4-week phases: early adoption (weeks 1 to 4) and late adoption (weeks 5 to 8). Participants in both groups will engage in pre-recorded exercise content. The AEP + SHC group may receive up to 12 health coaching calls. Machine learning will be used in Weeks 2, 6, and 10 to predict which AEP + HC participants should receive coaching calls for the next four weeks.

The proposed Sequential Multiple Assignment Randomized Trial (SMART) study seeks to develop an effective 32-week, resource-sensitive strategy to improve physical activity levels in people with mobility impairments. During the run-in period before the start of the intervention, interested individuals will consent to be part of the study. Once providing consent, participants will respond to a baseline survey packet through REDCap. Participants must also complete a welcome call and set up an online account. Additionally, during the run-in period, the research team will ship an exercise tracker device, and an exercise band for the participant to wear during the intervention. The participant will receive an orientation call to assist them with using the website, setting up their exercise tracking device, and linking the device to the website. After the run-in period, participants will be randomized into 1 of 2 groups: Asynchronous Exercise Program (AEP) and AEP + Smart Health Coaching (SHC). Finally, participants will be given access to the FitWithUs online platform, hosted on UAB servers, to access all the exercise content (exercise videos and articles). All participants will receive at least one new health and wellness article per week for eight weeks, and new exercise videos for 16 weeks. This intervention will be administered in 8 waves of ~33-34 participants each (pilot wave data excluded from analyses). The Adoption Phase will be split into two 4-week phases: early adoption (weeks 1 to 4) and late adoption (weeks 5 to 8). Participants in both groups will engage in pre-recorded exercise content. The AEP + SHC group may receive up to 12 health coaching calls. Machine learning will be used in Weeks 2, 6, and 10 to predict which AEP + HC participants should receive coaching calls for the next four weeks. At the end of the early adoption phase, the participant will complete a short set of questions (See week 4 questionnaire) the research team will classify participants in both groups into either a responder or a non-responder. If a participant is a responder, they will continue with their group assignment through the late adoption phase (AEP only or AEP + SHC). If the participant is a non-responder, they will be randomized a second time into 1 of 2 sub-groups: Live 1-on-1 training or Live group training for the late adoption phase. All live training will occur remotely through ZOOM. Participants in non-responder sub-groups will be asked to participate in their respective live training up to 3 times per week for weeks 5 to 8. This second randomization results in six possible intervention groups: 1) AEP only responder, 2) AEP + HC responder, 3) AEP non-responder + LAT_1-1, 4) AEP non-responder + LAT_GRP, 5) AEP + HC non-responder + LAT_1-1, 6) AEP + HC non-responder + LAT_GRP. Upon finishing the late adoption phase, all participants will complete another survey packet and a semi-structured interview (see interview guide), and receive AEP only for a 24-week maintenance phase (weeks 9-32). Upon completion of week 32, the participant will complete a final survey packet. Throughout the study, we will be collecting data from the participant's exercise tracker. These data include steps and minutes of activity/inactivity. During weeks 9 to 32, participants will have open access to the website and its library of exercise content. The research team will continue to collect activity data and website analytics (for example video watch minutes). Participants may receive a reminder call to complete surveys. We will use the following validated measures: [existing measures list unchanged].

ELIGIBILITY:
Eligible participants must meet the following criteria to be included: (1) live with a permanent physical disability that limits their mobility; (2) be 18 to 89 years of age; (3) have broadband internet access; (4) be able to speak and read English; and (5) be able to attend coaching and training sessions during the weekdays.

Participants are excluded from participation if they (1) possess significant visual acuity that prevents seeing a computer screen to follow a home exercise program; (2) have been regularly engaging in exercise for the previous 3 months; (3) are unable to use their arms and their legs at all to exercise; (4) are unsafe to exercise; (5) self-report that they are currently pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Fitbit: ongoing for 32 weeks; Godin: Baseline, week 8, week 16, and week 32
  The primary outcome is the change in physical activity (steps per day) from baseline to the end of the 32-week intervention.
  Participants wear Fitbit Inspire 3 trackers (Google LLC, Sacramento, CA) for continuous objective measurement, with data exported via the study dashboard.
  This is supplemented by the Godin Leisure-Time Exercise Questionnaire (GLETQ) at baseline, week-8 and week-16 for self-reported leisure-time activity in MET-minutes/week.

SECONDARY OUTCOMES:
Health information technology literacy | Baseline, week 8, week 16, and week 32
  The secondary outcome is health information technology literacy, measured by the eHealth Literacy Scale (eHEALS).
  The eHEALS is a validated 8-item questionnaire assessing participants' perceived skills in finding, evaluating, and applying online health information (scored 8-40).
  Assessments occur at baseline, week 8, week 16, and week 32 to track changes over the 32-week intervention.
Secondary Health Conditions | Baseline, week 8, week 16, and week 32
  The secondary outcome is secondary health conditions, assessed via National Institutes of Health Patient-Reported Outcome Measurement Information System (PROMIS) questionnaires.
  PROMIS measures include pain interference, fatigue, sleep disturbance, and quality of life, each on a T-score metric (mean 50, SD 10) for standardized comparison.
  Assessments occur at baseline, week 8, week 16, and week 32 to evaluate changes over the 32-week intervention.
Activity limitations | Baseline, week 8, week 16, and week 32
  The secondary outcome is activity limitations, measured by the Physical Functioning subscale of the 36-Item Short Form Survey (SF-36 PF).
  The SF-36 PF is a validated 10-item questionnaire assessing limitations in physical activities due to health problems (scored 0-100, higher scores indicate better functioning).
  Assessments occur at baseline, week 8, week 16, and week 32 to track changes over the 32-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mohanraj Thirumalai, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Wellness, Health and Research Facility, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Intervention landing page. — https://fitwithus.org/